CLINICAL TRIAL: NCT04581590
Title: Can Task Specificity and Baseline Outcomes Impact TDCS-linked Motor and Cognitive Training Gains in Parkinson's Disease? a Protocol for a Controlled, Double-blind, Randomized Multicentric Clinical Trial
Brief Title: The Impact TDCS-linked Motor and Cognitive Training Gains in Parkinson's Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Collaborators: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Suellen Andrade, Principal Investigator and Professor, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: tDCSparkinson
Record Dates: First submitted 2020-08-31; First posted 2020-10-09 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Parkinson Disease; Cognition Disorder; Motor Disorders
MeSH Terms: conditions — Parkinson Disease; Cognition Disorders; Motor Disorders | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: This is a sham-controlled, double-blind randomized multicentric clinical trial will analyze patients with a confirmed diagnosis of Parkinson disease who were subjected to tDCS associated with dual-task motor training and cognitive tranining
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active group (Active Comparator): In the group G1 will be administered: tDCS active + dual-task motor training + cognitive training.
  Interventions: Other: Cognitive training
- Sham group (Sham Comparator): In the group G2 will be administered: tDCS active + dual-task motor training
  Interventions: Other: Cognitive training

INTERVENTIONS:
Other: Cognitive training — Both groups will undergo the motor training where only the type of received electric current is varied (active or simulated sham type) associated cognitive training. The twelve sessions will be performed in three sessions per week for 30 minutes.
  Other Names: tDCS active

SUMMARY:
This study is a group controlled clinical trial. Parallel study, patients aged 40-70 years, with Parkinson disease. Twelve sessions, three times a week, for 30 minutes, simultaneously to the rehabilitation program. Training will consist of Transcranial Direct Current Stimulation linked dual-task exercises or dual-taks exercises with cognitive training, applied three times a week during four weeks. The investigators will used instruments: dual-task gait speed (Auditory Stroop Task ), executive function (Wisconsin Card Sorting Test , Auditory Stroop Test, Trail Making Test, Verbal Fluency Test and Montreal Cognitive Assessment), and, the objective is to examine task-dependency in enhancing the effects of tDCS-linked rehabilitation training on PD and the relationships between baseline outcomes in responders and non-responders to therapy.

DETAILED DESCRIPTION:
Background: Patients with Parkinson's disease have difficulty performing a dual-task, a condition present in everyday life. It is possible that strategies such as Transcranial Direct Current Stimulation can be associated with motor training enriched with dual-task and cognitive training to improve the performance of two concurrent tasks. It is currently unclear whether specific tasks and clinical conditions of PD patients have different results after the intervention. Therefore, the proposed randomized controlled trial will examine task-dependency in enhancing the effects of tDCS-linked rehabilitation training on PD and the relationships between baseline outcomes in responders and non-responders to therapy.

Discussion: This study will evaluate the effectiveness of an intervention protocol with transcranial direct current stimulation, dual-task training and cognitive training in patients with Parkinson's disease. The study will also highlight whether the clinical factors and variability between individuals that could interfere in the training of a specific task and influence the therapeutic effect.

ELIGIBILITY:
Inclusion Criteria:

* being diagnosed with idiopathic Parkinson's disease by a neurologist based on definitive evidence of responsiveness to levodopa at the start of the disease and the history of progressive hypokinesia with asymmetric onset. PD will be diagnosed based on Parkinson's Disease Society Brain Bank (PDSBB) criteria, as described in Hughes et al.
* age between 40 and 70 years, with no distinction for sex, schooling level or other sociodemographic characteristics
* disease staging between 1.5 and 3, according to the modified Hoehn and Yahr scale
* undergoing regular pharmacological treatment with levodopa (equivalent dose > 300mg) or taking antiparkinsonian medication such as anticholinergics, selegiline, dopamine agonists (amantadine) and COMT (catechol-O-methyl transferase) inhibitors
* score of more than 24 points on the Mini-Mental State Examination
* not exhibiting other associated neurological diseases and no musculoskeletal and/or cardiorespiratory changes that could compromise gait.

Exclusion Criteria:

* be diagnosis of atypical Parkinson's disease
* neuropsychiatric comorbidities; convulsions, metal clips and/or pacemaker; deep brain stimulation implant; history of epilepsy; neurosurgery; traumatic brain injury; alcohol abuse or drug dependency;
* associated diseases of the peripheral or central nervous system
* undergoing physical therapy at another location
* inability to walk 10 meters
* presence of important dyskinesia that prevents the participant from sitting in a chair
* abnormal and persistent increase in systemic blood pressure before or during training, after 3 measurements taken 5 minutes apart - Cut-off: systolic blood pressure ≥ 140 mm Hg and/or diastolic ≥ 90 mm Hg
* not understanding any of the training protocol stages
* chemical scalp treatment within the previous 30 days, and experiencing severe pain and/or discomfort that precludes performing the proposed activities.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
Changes dual-task gait speed by the Auditory Stroop Task | [Baseline, after 04 weeks]
  For this outcome, the Auditory Stroop Task participants will be asked to walk while listening to words spoken loudly and softly and indicate if the volume heard was loud or low, irrespective of the word pronounced.

SECONDARY OUTCOMES:
Changes in executive functions assessed by Wisconsin Card Sorting Test (WCST) | [Baseline, after 04 weeks]
  The Wisconsin Card Sorting Test (WCST) is a neuropsychological test of "set-shifting", i.e. the ability to display flexibility in the face of changing schedules of reinforcement. A number of stimulus cards are presented to the participant. The participant is told to match the cards, but not how to match; however, they are told whether a particular match is right or wrong. The original WCST used paper cards and was carried out with the experimenter on one side of the desk facing the participant on the other. The test takes approximately 12-20 minutes to carry out and generates a number of psychometric scores, including numbers, percentages, and percentiles of: categories achieved, trials, errors, and perseverative errors.
Changes in executive functions assessed by Trail Making Test (TMT) | [Baseline, after 04 weeks]
  The Trail Making Test (TMT) is a neuropsychological test of visual attention and task switching. It consists of two parts in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy.The test can provide information about visual search speed, scanning, speed of processing, mental flexibility, as well as executive functioning
Changes in executive functions assessed by Verbal Fluency Test | [Baseline, after 04 weeks]
  The Verbal Fluency Test are a kind of psychological test in which participants have to produce as many words as possible from a category in a given time (usually 60 seconds). This category can be semantic, including objects such as animals or fruits, or phonemic, including words beginning with a specified letter, such as p, for example
Changes in executive functions assessed by Montreal Cognitive Assessment (MoCA) | [Baseline, after 04 weeks]
  The Montreal Cognitive Assessment (MoCA) is a cognitive screening tool. MoCA is composed of eight cognitive domains, which are scored within a range of 0 to 30 points (higher scores indicate better function): short-term memory; visuospatial skills; executive function; verbal fluency; attention, concentration and working memory; language; sentence repetition; and spatiotemporal orientation.
Changes in motor functions assessed by Dynamic Gait Index (DGI) | [Baseline, after 04 weeks]
  The Dynamic Gait Index (DGI) assess gait, balance and fall risk. It evaluates not only usual steady-state walking, but also walking during more challenging tasks. A four-point ordinal scale, ranging from 0-3. "0" indicates the lowest level of function and "3" the highest level of function (total score = 24).
Changes in motor functions assessed by 10-meter walk test | [Baseline, after 04 weeks]
  The 10-meter walk test to estimate gait speed by recording the average time the patient takes to cover a distance of 10m in three attempts
Changes in motor functions assessed by Timed Up and Go (TUG) test | [Baseline, after 04 weeks]
  The Timed Up and Go (TUG) test to stand up from a chair at the command, walk 3 meters walk along a demarcated course, turn around and walk back to the chair, then sit down.
Changes in motor functions assessed by Kinematics of Gait | [Baseline, after 04 weeks]
  To analyze movement using the Qualisys Motion Capture System (Qualisys Medical AB, 411 13, Gothenburg, Sweden);
Changes in motor function assessed by the Unified Parkinson's Disease Rating Scale - Part III (UPDRS - III) | [Baseline, after 04 weeks]
  For this outcome, the Unified Parkinson's Disease Rating Scale - Part III will be used. Section III provides an overall score for movement-related functions and activities (tremor, stiffness, gait, alternating movements, among others). This section is made up of 33 items, which can range from zero (normal) to four (severe), with responses that are linked to commonly accepted clinical terms. The higher the score, the greater the impairment of motor function.
Changes in motor function assessed by Activities-specific balance confidence (ABC) scale | [Baseline, after 04 weeks]
  For this outcome, Activities-specific balance confidence (ABC) scale to measure the level of confidence in performing daily activities, in addition to identifying fear of falling and possible social isolation
Changes in sleep quality assessed by Parkinson's disease sleep scale-2 (PDSS-2) | Time Frame: [Baseline, after 04 weeks]
  The PDSS is a scale specifically designed to assess sleep quality in individuals with Parkinson's. The PDSS-2 consists of 15 questions rated according to five categories ranging from 0 (never) to 4 (very frequent). Its total score ranges from 0 (no disturbance) to 60 (maximum nighttime disturbance).
Changes in sleep quality assessed by Pittsburgh Sleep Quality Index (PSQI) | Time Frame: [Baseline, after 04 weeks]
  The Pittsburgh Sleep Quality Index (PSQI) is a widely used self-report questionnaire that assesses sleep quality over a one-month time interval. Each component score of the PSQI ranges from 0 to 3, with 3 indicating the greatest dysfunction or disturbance. The seven component scores are then summed to obtain a global PSQI score, which ranges from 0 to 21. Higher scores indicate poorer sleep quality, with a score greater than 5 suggesting significant sleep difficulties.
Changes in daytime sleepiness assessed by the Epworth Sleepiness Scale (ESS) | Time Frame: [Baseline, after 04 weeks]
  The ESS is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'.

CONTACTS AND LOCATIONS:
Overall Officials: Suellen Suellen Andrade, Principal Investigator — Federal University of Paraíba
Locations (1):
- Federal University of Paraíba, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Costa-Ribeiro A, Andrade SMMDS, Ferrer MLV, Silva OAPD, Salvador MLS, Smaili S, Lindquist ARR. Can Task Specificity Impact tDCS-Linked to Dual Task Training Gains in Parkinson's Disease? A Protocol for a Randomized Controlled Trial. Front Aging Neurosci. 2021 Jul 1;13:684689. doi: 10.3389/fnagi.2021.684689. eCollection 2021. PMID 34276344